CLINICAL TRIAL: NCT03833089
Title: Arrhythmia Prevention in High Risk Cardiovascular Patients Using Targeted Potassium Levels
Brief Title: Targeted Potassium Levels for Prevention of ICD Therapy
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Christian Joens, Staff Cardiologist, Electrophysiology, Principal investigator, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3589
Record Dates: First submitted 2019-02-01; First posted 2019-02-06 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Ventricular Arrhythmias and Cardiac Arrest; Implantable Defibrillator User; Hypokalemia; Hyperkalemia; Ventricular Tachycardia; Atrial Fibrillation
MeSH Terms: conditions — Heart Arrest; Hypokalemia; Hyperkalemia; Tachycardia, Ventricular; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): ICD recipients in optimal Medical treatment as per guidelines according to their comorbidity
- Targeted serum potassium levels (Experimental): ICD recipients recipients in optimal Medical treatment as per guidelines according to their comorbidity. In addition to guideline recommended treatment, this cohort will be treated to increase serum potassium levels to 4.5-5.0 mEq/L.
  Interventions: Combination Product: Targeted serum potassium level

INTERVENTIONS:
Combination Product: Targeted serum potassium level — In the following order, following advices end prescriptions will be provided: 1) Potassium rich dietary advice, 2) Mineralocorticoid receptor antagonists, 3) Potassium supplementation,
  Arms: Targeted serum potassium levels

SUMMARY:
This study evaluates whether a rigorously controlled high-normal level of serum-potassium (4.5-5.0 mEq/L) using dietary recommendations, potassium supplements and mineralocorticoid receptor antagonists will results in a lower incidence of cardiac arrhythmias in patients with an ICD. Patients will be randomized to this treatment or a control arm, where patients will receive usual guideline recommended follow-up.

DETAILED DESCRIPTION:
There is solid evidence that potassium-sparing drugs increase survival and ameliorates symptoms in heart failure patients and post-hoc studies have suggested that high-normal levels of blood potassium levels (p-K) markedly decreases the risk of malignant arrhythmias in cardiovascular patients.

This trial will randomize patients implanted with implantable cardioverter defibrillators (ICDs), who remain at high risk of life-threatening cardiac arrhythmias, to a standard therapy or standard therapy plus a regimen to keep high-normal p-K levels. The study will enroll 1,000 patients from the outpatient pacemaker clinics at Rigshospitalet and Gentofte hospital. Using a planned regime to increase p-K using inexpensive drugs and potassium supplements, the patients enrolled and followed with regular controls as well as continuous monitoring using existing home monitoring systems over a period of 4 years for the primary endpoint of appropriate ICD therapy and all cause mortality. Including analysis, the trial will be running for 5 years

ELIGIBILITY:
Inclusion Criteria:

* Implantable cardioverter defibrillator (ICD) or cardiac resynchronization pacemaker with ICD (CRT-D).
* Age >18 years

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) <30 ml/h
* Pregnancy
* Lack of ability to understand and sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-05-09 (Estimated); Study Completion 2035-04-01 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of ECG documented ventricular tachycardia, appropriate ICD therapy, hospitalization > 24 hours due to arrhythmias and/or heart failure leading to a change in treatment and all cause mortality | Total 291 events, expected 6 years
  A combination of:
  * ECG documented ventricular tachycardia > 125 bpm lasting > 30 seconds
  * Any appropriate ICD therapy as documented by the ICD or ECG
  * Any unplanned hospitalizations > 24 hours due to arrhythmias and/or heart failure leading to a change in treatment, e.g., administration of new drugs, or change in doses of already prescribed drugs or invasive or non-invasive treatment.
  * All-cause mortality
  The time period with regards to the Time-to-Event Outcome Measures starts with the randomization of the patient.
  ECG documented tachycardia from ECGs or ICD interrogations will be obtained from hospitalizations or outpatients clinic visits via electronic records after patient consent. Information of ventricular tachyarrhythmia therapy will be obtained from home monitoring systems or interrogation of the ICD devices during in-clinic visits.
  Mortality will be obtained from danish electronic hospital files or the danish death registry.

SECONDARY OUTCOMES:
Time to first incidence of supraventricular arrhythmias as documented by ECG or the ICD | 6 years
  Any supraventricular tahcycardia documented on ECG, telemetry or as monitored/treated event on the ICD
Proportion of patients experiencing <92 % CRT-pacing for > 2 weeks (only CRT-D patients) | 6 years
  CRT-D home monitoring systems allow temporal evaluation of percentage of CRT pacing.
Time to first hospitalization for heart failure | 6 years
  Hospitalization with symptoms of heart failure and with a diagnosis of heart failure where treatment with i.v. diuretics was initiated.
Time to first hospitalization for cardiac arrhythmias | 6 years
  Hospitalization were records indicate that supraventricular or ventricular arrhythmias were implicated in the cause of the hospitalization
Time to hospitalization for electrolyte disturbances or kidney failure | 6 years
  Hospitalization were records indicate that kidney failure or disturbances in the potassium or sodium plasma leves were implicated in the cause of the hospitalization
First occurrence of appropriate ICD therapy for ventricular tachycardia or ventricular fibrillation irrespective of outcome. | 6 years
  Ventricular tachy-arrhythmia therapy, which will be obtained from home monitoring systems or interrogation of the ICD devices during in-clinic visits. All ICD therapy is routinely adjudicated as appropriate or in-appropriate by electrophysiologists at the study sites.
Time to first occurence of inappropriate ICD therapy | 6 years
  Any cause of inappropriate shock including atrial fibrillation, other supraventricular arrhythmias, ICD lead problems etc.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Joens, MD, PhD, Principal Investigator — Dept of Cardiology, Rigshospitalet, Denmark; Niels Risum, MD, PhD, Study Chair — Dept of Cardiology, Rigshospitalet, Denmark; Henning Bundgaard, Prof., DMSc, Study Chair — Dept of Cardiology, Rigshospitalet, Denmark
Locations (3):
- Denmark (3):
  - Gentofte University Hospital, Gentofte Municipality, Hellerup
  - Roskilde University Hospital, Roskilde, Region Sjælland
  - Rigshospitalet, Copenhagen

REFERENCES:
- [Derived] Jons C, Zheng C, Winslow UCG, Danielsen EM, Sakthivel T, Frandsen EA, Saffi H, Vakilzadeh-Hashemi SS, Haugan KJ, Bruun NE, Iversen KK, Bosselmann HS, Risum N, Bundgaard H; POTCAST Study Group. Increasing the Potassium Level in Patients at High Risk for Ventricular Arrhythmias. N Engl J Med. 2025 Nov 20;393(20):1979-1989. doi: 10.1056/NEJMoa2509542. Epub 2025 Aug 29. PMID 40879429
- [Derived] Winslow U, Sakthivel T, Zheng C, Bosselmann H, Haugan K, Bruun N, Larroude C, Iversen K, Saffi H, Frandsen E, Oturai P, Jensen HJ, Vinther M, Risum N, Bundgaard H, Jons C. Treatment-induced increase in total body potassium in patients at high risk of ventricular arrhythmias; a randomized POTCAST substudy. PLoS One. 2023 Jul 19;18(7):e0288756. doi: 10.1371/journal.pone.0288756. eCollection 2023. PMID 37467227

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT03833089/Prot_SAP_001.pdf